CLINICAL TRIAL: NCT00420134
Title: A Phase One/Two Clinical Trial on the Use of Autograft Mesenchymal Stem Cells Differentiated Into Progenitor of Hepatocytes for the Salvage Treatment of Patients With End-stage Liver Disease
Brief Title: Improvement of Liver Function in Liver Cirrhosis Patients After Autologous Mesenchymal Stem Cell Injection:a Phase I-II Clinical Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Tarbiat Modarres University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 348
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Liver Failure; Cirrhosis
Keywords: mesenchymal stem cell; end stage liver disease; Cirrhosis; stem cell therapy
MeSH Terms: conditions — Liver Failure; Fibrosis; End Stage Liver Disease

INTERVENTIONS:
Procedure: injection of progenitor of hepatocyte drived from Mesenchymal stem cell

SUMMARY:
The methods for separation of mesenchymal stem cell were established in 2001. These cells can differentiate to osteocytes, hepatocytes, chondrocytes, myocytes and etc,. In this study the investigators try to separate mesenchymal stem cell from end stage liver disease, then these cells will be differentiated to progenitor of hepatocytes, finally , the investigators injected these cells into portal vein under ultrasound guide. The investigators determine the effects of injected cells in reestablishment of liver function.

ELIGIBILITY:
Inclusion criteria:

* MELD score of at least 10
* Patent portal vein on color Doppler examination of the liver
* Normal alpha-feto protein serum levels
* Age more than 18
* Filling inform consent by patients and first degree family members

Exclusion criteria:

* Any evidence of hepatocellular carcinoma on liver ultrasound studies
* Patients want to exclude from study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Liver function test
MELD score

SECONDARY OUTCOMES:
Cirrhosis mortality after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Reza Zali, MD, Study Chair — Research center of Gastroenterology and Liver Disease; Pedram Kharaziha, MD, Principal Investigator — Research Center for Gastroenterology and Liver Diseases
Locations (2):
- Iran (2):
  - Research Center for Gastroenterology and Liver Diseases, Tehran, Tehran Province
  - Research center of Gastroenterology and Liver Disease, Tehran, Tehran Province